CLINICAL TRIAL: NCT03929107
Title: Interleukin-7 and Chemokine (C-C Motif) -Ligand 19-expressing CD19-CAR-T for Refractory/Relapsed B Cell Lymphoma
Brief Title: Interleukin-7 and Chemokine (C-C Motif) Ligand 19-expressing CD19-CAR-T for Refractory/Relapsed B Cell Lymphoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenbin Qian (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Sponsor-Investigator, Wenbin Qian, Doctor, Professor, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lymphoma center Q003
Record Dates: First submitted 2019-04-22; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: B Cell Lymphoma
Keywords: interleukin 7, Chemokine (C-C Motif) Ligand 19, CAR-T
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Interleukin-7; Chemokines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): In this group, patients will be treated with Interleukin-7 and Chemokine (C-C Motif) Ligand 19-expressing CD19-CAR-T, and the safety and efficacy will be evaluated.
  Interventions: Biological: Interleukin-7 and Chemokine (C-C Motif) Ligand 19-expressing CD19-CAR-T cells

INTERVENTIONS:
Biological: Interleukin-7 and Chemokine (C-C Motif) Ligand 19-expressing CD19-CAR-T cells — patient's T cells were seperated and engineered into Interleukin-7 and Chemokine (C-C Motif) Ligand 19-expressing CD19-CAR-T cells, and retransfused into the patient for treatment of their B cell lymphoma.

SUMMARY:
It's a single arm, open label prospective study, in which the safety and efficacy of Interleukin-7 and Chemokine (C-C Motif) Ligand 19-expressing CD19-CAR-T therapy are evaluated in refractory/relapsed B cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old, male or female;
* 2. ECOG 0-3, for patients with ECOG=4, if ECOG reach 0-3 after bridging treatment with ibrutinib, they are also considered to fit this criteria;
* 3. Histologically diagnosed as B cell non-Hodgkin's lymphoma (NHL)(according to WHO 2008 criteria), including DLBCL-NOS, primary mediastinal B cell lymphoma (PMBCL) mantel cell lymphoma (MCL), transformed follicular lymphoma (TFL) and other transformed B cell NHL;
* 4. CD19 positive (by immuno-histology or flowcytometry) [for DLBCL/PMBCL/TFL patients, negative CD19 immuno-histology results also acceptable];
* 5. Definition of relapsed and refractory disease: 1) refractory DLBCL should fit one of the following: ①complete remission NOT achieved after 2nd line treatment; ②progression of disease during treatment; ③duration of stable disease <6 months; ④ disease progress or relapse within 12 months of autologous stem cell transplantation.

  2) definition of refractory/relapsed disease for CLL and other indolent B cell NHL, should fit one of the following: ① failed or relapsed after 2nd therapy (Rituximab must be included) and being unable to accept ibrutinib treatment due to various reasons; ② non-responsive or intolerable to ibrutinib as 2nd line treatment; 3) refractory or relapsed MCL should fit one of the following: ① complete remission not achieved after 2nd line treatment; ② disease progression during treatment; ③duration of stable disease ≤6 months; ④disease progress or relapse within 12 months of autologous stem cell transplantation.
* 6. Previous treatment of aggressive B lymphomas must include Rituximab and anthracyclines;
* 7. Patients should have at least one measurable disease focus, with the longitudinal diameter ≥1.5cm, or any extra-nodal focus with the longitudinal diameter ≥1.0cm, with PET/CT positive results;
* 8. Blood routine test, absolute neutrophil count≥1000/ul、platelet count≥45000/ul；
* 9. Cardiac, hepatic and renal function: Creatinin <1.5 times of normal maximum；ALT/AST level <2.5 times of the maximum of normal range; total bilirubin<1.5 times of ULN；cardiac ejection fraction≥ 50%;
* 10. Patients should have the ability to fully understand contents of the written consent and be willing to sign the written consent;
* 11. Fertile patients should agree to take contraceptive measures during the process of this trial.

Exclusion Criteria:

* 1. History of other malignant tumor;
* 2. History of autologous stem cell transplantation within 6 weeks prior to enrollment;
* 3. Received CAR-T therapy within 3 months prior to enrollment;
* 4. Received cytotoxic medicine or glucocorticoids or other targeted-therapy medicine (except for ibrutinib) within 2 weeks prior to T cell collection;
* 5. With active autoimmune disease;
* 6. With active infection;
* 7. With HIV infection, or uncontrolled HBV/HCV/syphilis infection;
* 8. With known central nervous system lymphoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | at the time point 3 months after CAR-T cell transfusion
  complete remission rate after treated by CAR-T therapy
adverse events | from the date of the start of treatment to 24 months after last patient's enrollment
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

SECONDARY OUTCOMES:
progression free surviva | from the day of treatment to the date of first documented progression，up to 24 months after the last patient's enrollment
  from date of inclusion to date of progression, relapse, or death from any cause
overall survival | from the day of treatment to the date of first documented progression，up to 24 months after the last patient's enrollment
  from the date of inclusion to date of death, irrespective of cause
duration of the CAR-T cells in the patients | from the date of re-transfusison to 24 months after last patient's enrollment
  time from re-transfusion to date when the modified T cells become non-detectable.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, MD，PhD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China